CLINICAL TRIAL: NCT07169097
Title: Study of the Pharmacokinetics of Ceftriaxone in Urinary Tract Infections in the Emergency Department
Brief Title: Study of the Pharmacokinetics of Ceftriaxone
Acronym: Etude PC-IUU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/212/OB; 2023-A02238-37 (Other: ANSM)
Record Dates: First submitted 2025-09-01; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Urinary Infections
Keywords: antibiotic; cephalosporin; therapeutic target; pharmacokinetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 4 mL dry tube and a 4 mL heparinized tube will be collected for the determination of total and free ceftriaxone, albumin and bilirubin concentration in the blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: free ceftriaxone concentration dosage — The proportion of patients with UTI for whom the time spent with a free ceftriaxone concentration above 1x MIC is 100% will be determined by calculating the ratio of the total number of patients meeting this criterion to the total number of patients included. Plasma ceftriaxone dosages will be integrated into a structural model from the scientific literature using the MonolixSuite 2023R1® package (Lixoft - Saclay) including a modeling module (Monolix) and a simulation module (Simulx). T. Individual pharmacokinetic parameters will be determined by Bayesian estimation by integrating the dosage performed in the protocol.

SUMMARY:
Urinary tract infections (UTIs) are the leading cause of community-acquired bacterial infections in adults. They are a common reason for admission to the Emergency Department (ED), particularly when pyelonephritis is suspected. The main bacteria responsible for UTIs are Enterobacteriaceae, with Escherichia coli being the main cause, found in more than 90% of cases. The French guidelines of the SPLIF (French-Speaking Infectious Pathology Society) recommend the probabilistic use of a 3rd generation cephalosporin or a fluoroquinolone. Ceftriaxone is often chosen over cefotaxime because it can be injected only once a day, which simplifies its administration in overcrowded emergency departments. There are currently no SPLIF recommendations regarding the dosage of ceftriaxone to be administered. The IDSA (Infectious Diseases Society of America) suggests a single dosage of 1 gram/day. Ceftriaxone is a 3rd generation cephalosporin antibiotic in the β-lactam class. Its mechanism of action is based on the inhibition of bacterial cell wall synthesis. Due to its broad spectrum against Gram-positive and Gram-negative aerobic bacteria and also some anaerobic germs, ceftriaxone is a commonly prescribed antibiotic in emergency departments (Therapeutic Guidelines Limited, Melbourne, 2014; Kumar et al., 2009) because of its broad indications: neuromeningeal infections, intra-abdominal infections and urinary tract infections (UTIs). Since most UTIs requiring hospitalization do not require intensive care, the optimal dosage of ceftriaxone in this context remains to be determined. Indeed, patients in emergency departments are on average less serious, without sepsis or septic shock, and therefore with probably different pharmacokinetic parameters.

DETAILED DESCRIPTION:
While PK data in healthy volunteers support a single dose of ceftriaxone 1 gram/day, those from intensive care patients support 2 or even 4 grams/day. Febrile UTIs are a heterogeneous group of patients ranging from simple acute pyelonephritis in young women with no history to complex urinary tract infection in malnourished elderly patients and male urinary tract infection in elderly patients with benign prostatic hyperplasia. The present project therefore aims to evaluate whether a single dose of 1 g of ceftriaxone is sufficient to achieve the therapeutic target in all patients suffering from febrile UTI without septic shock or whether certain situations would justify a dosage adjustment. To this end, patients presenting a clinical and biological picture of UTI and having received ceftriaxone administration will be offered inclusion in this protocol. A 4 mL dry tube and a 4 mL heparinized tube will be collected for the determination of total and free ceftriaxone, albumin, and bilirubin concentrations. These samples will be added to the assessment performed as part of routine care within 24 hours of the first ceftriaxone injection. This study will calculate the probability of reaching the therapeutic target in patients treated with ceftriaxone for UTI without septic shock. Depending on the results, this study could allow the proposal of a personalized dosage of ceftriaxone for each patient suffering from urinary tract infection based on their clinical and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age
* Requiring hospitalization at Rouen University Hospital
* Clinical diagnosis of urinary tract infection requiring ceftriaxone antibiotic therapy
* Prescription of 1g IV ceftriaxone
* Venipuncture for laboratory testing as part of the prescribed treatment within 24 hours of the first ceftriaxone injection
* Patient has read and understood the information letter and given oral consent to participate in the study

Exclusion Criteria:

* Minor patient
* Patient hospitalized in an intensive care unit
* Patient with septic shock
* Chronic dialysis or indication for emergency renal replacement therapy (ERP)
* Prescription of a dosage other than 1g intravenously per 24 hours
* Patient having received more than one injection of 1g ceftriaxone
* Pregnant, parturient, or breastfeeding woman
* Person deprived of liberty by an administrative or judicial decision
* Person placed under judicial protection, guardianship, or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (>18 years) with clinical diagnosis of urinary tract infection requiring antibiotic therapy with ceftriaxone at a dose of 1g/24h intravenously (IV).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with urinary tract infection (UTI) for whom the time spent with a free ceftriaxone concentration | within 24 hours after enrollment visit
  To determine the proportion of patients with UTI for whom the time spent with a free ceftriaxone concentration above 1x MIC is 100% (fT > 1x MIC = 100%). The primary objective will be evaluated by simulation using a two-compartment population pharmacokinetic model whose initial parameters will be set in accordance with the scientific literature. The residual concentration of free ceftriaxone will be used and compared to the critical concentration threshold of ceftriaxone for each pathogen defined by EUCAST (European Committee on Antimicrobial Susceptibility Testing).

SECONDARY OUTCOMES:
Determine the probability of reaching the efficiency threshold fT > 1x MIC = 100% for MICs varying from 0.25 to 32 mg/L | within 24 hours after enrollment visit
  For beta-lactams (BL) such as ceftriaxone, this is the fraction of time, fT, (expressed as a percentage between doses) where the free concentration of the antibiotic is above the minimum inhibitory concentration or MIC (%ƒT>MIC). - The probability of reaching the efficacy threshold fT > 1x MIC = 100% will be assessed using PTA (probability of target attainment) curves. Simulations will be performed using the pharmacokinetic model with different dosages and according to different MICs (from 0 to 32 mg/L).
Determine a mathematical function allowing the free plasma fraction of ceftriaxone to be extrapolated from the total ceftriaxone concentration | within 24 hours after enrollment visit
  The relationship between the free and total form of plasma ceftriaxone will be studied according to a linear binding model
Describe the microbial epidemiology of UTIs in the Emergency Department (ED) | within 24 hours after enrollment visit
  The microbial epidemiology of UTIs in the ED will be assessed by microbiological analysis of the ECBU of included patients collected retrospectively.
Determine the impact of clinical-biological variables on the pharmacokinetic profile of ceftriaxone (weight) | within 24 hours after enrollment visit
  The weight will be that measured from the patient. This variable will be analyzed centered on the mean with and without logarithmic conversion.
Determine the impact of clinical-biological variables on the pharmacokinetic profile of ceftriaxone (albuminemia) | within 24 hours after enrollment visit
  The dosages of albuminemia will be carried out using samples taken as part of the study. The variable will be analyzed centered on the mean with and without logarithmic conversion.
Determine the impact of clinical-biological variables on the pharmacokinetic profile of ceftriaxone (bilirubinemia) | within 24 hours after enrollment visit
  The dosages of bilirubinemia will be carried out using samples taken as part of the study. The variable will be analyzed centered on the mean with and without logarithmic conversion.
Determine the impact of clinical-biological variables on the pharmacokinetic profile of ceftriaxone (creatinineemia) | within 24 hours after enrollment visit
  The dosages of creatinineemia will be carried out using samples taken as part of the study. The variable will be analyzed centered on the mean with and without logarithmic conversion.
Determine a mathematical function allowing the free plasma fraction of ceftriaxone to be extrapolated from the total ceftriaxone concentration | within 24 hours after enrollment visit
  The relationship between the free and total form of plasma ceftriaxone will be studied according to an empirical saturation model
Determine a mathematical function allowing the free plasma fraction of ceftriaxone to be extrapolated from the total ceftriaxone concentration | within 24 hours after enrollment visit
  The relationship between the free and total form of plasma ceftriaxone will be studied according to different in vivo saturation models

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.